CLINICAL TRIAL: NCT06294158
Title: Light and Noise: Objectively Assessing Environmental Risk Factors for Delirium in the ICU
Acronym: LANYARD-ICU
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: LANYARD-ICU-1.1
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Delirium; Critical Illness
Keywords: Delirium; Critical Illness; Light; Noise
MeSH Terms: conditions — Delirium; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation Cohort: Adult patients (age ≥ 18 years) admitted to to participating Intensive Care Units with an expected (further) stay in participating Intensive Care Unit ≥ 48 hours who are not (currently) deeply sedated (RASS ≥ -3) and are not already in delirium (CAM-ICU positive), do not require environmental modification due to treatment necessities (e.g., burns care), and do not have advanced directives or treatment limitation orders in place, in whom environmental light and noise are measured.
  Interventions: Other: Brightness measurement; Other: Sound level measurement

INTERVENTIONS:
Other: Brightness measurement — Measurement of ambience brightness using lux meters
Other: Sound level measurement — Measurement of ambience sound levels using sound level meters

SUMMARY:
Recognition of delirium as a medical entity with relevance to both morbidity and mortality, especially in critically ill patients, is a relatively recent development. However, research into delirium prevention and treatment is now in focus of scientific efforts internationally.

Knowledge of intensive care unit (ICU) environment as a potential modifiable risk factor for delirium is insufficient to this date. This study thus seeks to evaluate, whether potentially modifiable environmental factors, such as noise or dazzling, are associated with development of delirium. Knowledge derived from this investigation could change both the process of care provision in intensive care units as well as the design of ICUs in general in the future.

This project is planned to be carried out as an observational pilot study at three perioperative ICUs at the University Medical Centre Graz. Adult patients shall be screened for inclusion, if not deeply sedated. Suitable patients shall be included into the study after written informed consent or deferred consent if they can be expected to remain in the ICU for at least another two days, if they are not already in delirium, if the ICU environment is not actively modified for therapeutic reasons and if no treatment limitations are in place. Over a study duration of one year, 250 to 300 patients are expected to be enrolled into the study. Of those, 60 to 120 patients are likely to develop delirium.

Baseline data known to be of relevance for outcome prediction in critically ill patients and factors known to predispose for development of delirium during ICU and hospital stay will be collected. Study equipment will be deployed to measure noise levels and illumination repeatedly over the day. Daily assessments for delirium using the Confusion Assessment Method in Intensive Care Units (CAM-ICU) will be performed. Vital status, physiologic parameters and parameters of ongoing treatment will concomitantly be documented on a daily basis.

Data on light and noise levels are then to be unified with parameters of physiology and treatment, vital status, and results of daily assessments for delirium. Statistical analysis using methods of descriptive and comparative statistics as well as both unadjusted and adjusted logistic regression analysis will be performed to identify factors significantly associated with the development of delirium (i.e., risk factors).

DETAILED DESCRIPTION:
Delirium - derived from the word lira, Latin for furrow - literally means "to get off track". Historically, signs and symptoms of delirium have been taunted as "insanity". Recognition of delirium as a medical entity with relevance to both morbidity and mortality, especially in in critically ill patients, is a relatively recent development. However, research into delirium, its prevention and treatment, is now in focus of scientific efforts by epidemiologic researchers and international societies alike.

Delirium now is a medical condition both recognised in current versions of the International Classification of Diseases (ICD-10) and the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). It is characterised by some disturbance in attention and awareness, acute onset and at least one additional disturbance in memory, orientation, language, visuospatial ability or perception, which cannot better be explained by another neurocognitive disorder and when there is evidence that the disturbances are a "direct physiological consequence" of another medical condition, substance intoxication or withdrawal, toxin, or various combinations of causes.

While historically sometimes regarded as an inalterable consequence of disease, delirium has been recognised as a significant contributor to both morbidity and even mortality in hospitalised patients, especially in critically ill individuals who require intensive care. Several risk factors for the development of delirium in intensive care units have been identified previously. However, many of these are factors not modifiable by caregivers (e.g., advanced age, frailty, pre-existing cognitive impairment, smoking, alcohol consumption, previous isolation, etc.) While some aspects of environment and interventions (especially endotracheal intubation, use of physical restraints and sedation with benzodiazepines, postoperative pain) have been found to be strongly associated with the development of delirium, assessment of the ICU environment itself as a potential modifiable risk factor is insufficient to this date.

Intensive care is known to be associated with high noise levels; attempts to reduce this noise pollution or provide protection from it may be worthwhile interventions to reduce delirium incidence. However, despite first attempts to establish associations between noise levels and delirium occurrence, no target values for possible future interventions have been established yet.

This study seeks to evaluate, whether potentially modifiable environmental factors in intensive care units, such as disturbances by noise or dazzling by light are associated with the development of delirium in critically ill patients. Knowledge derived from this investigation could change both the process of care provision in intensive care units as well as the design of ICUs in general in the future. Such changes could potentially improve outcomes, which would be much desired progress in delirium care, where both non-pharmacologic and pharmacologic therapeutic approaches have not convincingly been shown to be of benefit.

ELIGIBILITY:
Inclusion Criteria

* Adult patients (age ≥ 18 years)
* Admission to participating Intensive Care Unit
* Expected (further) stay in participating Intensive Care Unit ≥ 48 hours
* Not (currently) deeply sedated (RASS ≥ -3) Exclusion Criteria
* Patient already in delirium (CAM-ICU positive)
* Environmental modification due to treatment necessities (e.g., burns care)
* Advanced directives / Treatment limitation
* Current inclusion in other (interventional) trial
* Documented patient refusal in advance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients shall be included into the study if they can be expected to remain in the ICU for at least another two days, if they are not yet in delirium, if the ICU environment is not actively modified for therapeutic reasons (e.g., in the treatment of burns patients), if no treatment limitations are in place and if the patient can provide written informed consent. In those patients, who cannot provide informed consent upon recruitment due to their current illness or injury, consent by patients or their representatives shall be sought if and once they regain capacity (deferred consent).
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Delirium | 7 days
  Development of delirium, i.e., positive CAM-ICU examination

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Graz, Dept. of Anaesthesiology and Intensive Care Medicine, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided